CLINICAL TRIAL: NCT02568722
Title: STandard Versus Accelerated Initiation of Renal Replacement Therapy in Acute Kidney Injury (STARRT-AKI): A Multi-Centre, Randomized, Controlled Trial (Principal Trial)
Brief Title: Standard vs. Accelerated Initiation of RRT in Acute Kidney Injury (STARRT-AKI: Principal Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); National Health and Medical Research Council, Australia (Other); Baxter Healthcare Corporation (Industry); The George Institute (Other); National Institute for Health Research, United Kingdom (Other Government); Medical Research Institute of New Zealand (Other); Health Research Council, New Zealand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STARRT-AKI: Principal Trial
Record Dates: First submitted 2015-09-29; First posted 2015-10-06 (Estimated); Results first posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-07

CONDITIONS: Acute Kidney Injury
Keywords: Renal replacement therapy; Acute kidney injury; Dialysis; Hemodialysis; Critical illness
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard RRT initiation (Active Comparator): RRT initiation will be guided by the presence of one or more clinical indications. Even in the absence of one of these indications, RRT may be commenced at the discretion of the treating physician.
  Interventions: Other: Standard RRT initiation
- Accelerated RRT initiation (Experimental): A dialysis catheter will be placed and RRT initiated as soon as possible and within 12 hours of the patient meeting the eligibility criteria.
  Interventions: Other: Accelerated RRT initiation

INTERVENTIONS:
Other: Standard RRT initiation — In the absence of kidney function recovery, the initiation of RRT will be permitted if one of the following develops:
  serum potassium ≥ 6.0 mmol/L; pH ≤ 7.20 or serum bicarbonate ≤ 12 mmol/L; evidence of severe respiratory failure, based on a PaO2/FiO2 ≤ 200 and clinical perception of volume overload; and/or persistent AKI > 72 hours following the time of randomization.
  Arms: Standard RRT initiation
Other: Accelerated RRT initiation — A dialysis catheter will be placed and RRT initiated as soon as possible and within 12 hours of eligibility. This 12 hour window includes the time needed to obtain consent.
  Arms: Accelerated RRT initiation

SUMMARY:
The objectives of this trial are to determine whether, in critically ill patients with severe acute kidney injury (AKI), randomization to accelerated initiation of renal replacement therapy (RRT), compared to standard initiation, leads to:

1. Improved survival (primary outcome); and
2. Recovery of kidney function (principal secondary outcome), defined as independence from RRT at 90 days

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common and devastating complication of critical illness. Once AKI is established, treatment is largely supportive and no intervention has been found to restore kidney function or improve overall survival. Renal replacement therapy (RRT), usually in the form of hemodialysis, is frequently needed to manage patients with severe AKI. Such patients have an in-hospital mortality that consistently exceeds 50% with delays in RRT initiation implicated as a possible contributor. A recent meta-analysis suggested that earlier initiation of RRT may improve survival, but this is based on data derived overwhelmingly from observational studies. The investigators recently completed a multi-centre randomized controlled pilot trial that confirmed the feasibility of allocating patients to two different strategies of RRT initiation. Patient recruitment and follow-up, as well as patient safety, were successfully demonstrated during the pilot phase of this research program. The optimal timing of RRT initiation is an existing knowledge gap and a clear priority for investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Admission to an intensive care unit (ICU)
3. Evidence of kidney dysfunction [serum creatinine ≥100 µmol/L (women) and ≥ 130 µmol/L (men)]
4. Evidence of severe AKI defined by at least 1 of the following 3 criteria:

   i) ≥ 2-fold increase in serum creatinine from a known pre-morbid baseline or during the current hospitalization; OR ii) Achievement of a serum creatinine ≥ 354 µmol/L with evidence of a minimum increase of 27 µmol/L from pre-morbid baseline or during the current hospitalization; OR iii) Urine output < 6.0 mL/kg over the preceding 12 hours

Exclusion Criteria:

1. Serum potassium > 5.5 mmol/L
2. Serum bicarbonate < 15 mmol/L
3. Presence of a drug overdose that necessitates initiation of RRT
4. Lack of commitment to ongoing life support (including RRT)
5. Any RRT within the previous 2 months (either acute or chronic RRT)
6. Kidney transplant within the past 365 days
7. Known pre-hospitalization advanced chronic kidney disease, defined by an estimated glomerular filtration rate < 20 mL/min/1.73 m2
8. Presence or clinical suspicion of renal obstruction, rapidly progressive glomerulonephritis, vasculitis, thrombotic microangiopathy or acute interstitial nephritis
9. Clinician(s) caring for patient believe(s) that immediate RRT is mandated
10. Clinician(s) caring for patient believe(s) that deferral of RRT initiation is mandated

    * at their discretion, clinicians may administer a bolus of intravenous furosemide (ie, "furosemide stress test") and evaluate the subsequent urine output to help guide decision making regarding the likelihood of AKI progression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3019 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Wald, MDCM MPH, Principal Investigator — Unity Health Toronto; Sean M Bagshaw, MD MSc, Principal Investigator — University of Alberta
Locations (105):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida, Gainesville, Florida
  - University of Kentucy, Lexington, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
- Australia (16):
  - Ballarat Hospital, Ballarat
  - Flinder Medical Centre, Bedford Park
  - Bendigo Hospital, Bendigo
  - Eastern Hospital (Box Hill and Maroondah Hospital), Box Hill
  - Concord Hospital, Concord
  - The Northern Hospital, Epping
  - Geelong Hospital, Geelong
  - Austin Hospital, Heidelberg
  - Nepean Hospital, Kingswood
  - The Alfred Hospital, Melbourne
  - Nambour General Hospital, Nambour
  - Western Health (Footscray Hospital & Sunshine Hospital), St Albans
  - St. Vincent's Hospital, Sydney
  - Royal North Shore Hospital, Sydney
  - Royal Prince Alfred Hospital, Sydney
  - Princess Alexandra Hospital, Woolloongabba
- Austria (3):
  - Medical University Graz, Graz
  - Medical University Innsbruck, Innsbruck
  - Vienna General Hospital, Vienna
- Belgium (2):
  - Antwerp University Hospital, Edegem
  - Ghent University Hospital, Ghent
- Hospital de Clínicas de Porto Alegre - Rio Grande do Sul, Rio Branco, Brazil
- Canada (42):
  - Peter Lougheed Centre, Calgary, Alberta
  - Foothills Hospital, Calgary, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Red Deer Regional Hospital, Red Deer, Alberta
  - Sturgeon Community Hospital, St. Albert, Alberta
  - Surrey Memorial Hospital, Fraser Health, Surrey, British Columbia
  - St. Paul's Hospital - Providence Health Care, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - Health Sciences North, Greater Sudbury, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, University Hospital, London, Ontario
  - London Health Sciences Centre, Victoria Hospital, London, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Trillium Health Partners - Mississauga Hospital, Mississauga, Ontario
  - Lakeridge Health, Oshawa, Ontario
  - The Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Centre hospitalier de l'université de Montréal (Notre Dame), Montreal, Quebec
  - Centre hospitalier de l'université de Montréal (St. Luc), Montreal, Quebec
  - CHUM - Hôtel Dieu Montreal, Montreal, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec- Université Laval (IUCPQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Quebec (CHUQ), Québec, Quebec
  - Centre Hôspitalier universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec
  - Centre de sante et de services sociaux de Trois-Rivieres (CIUSSS MCQ), Trois-Rivières, Quebec
  - Regina Qu'Appelle Health Region, Saskatoon, Saskatchewan
- China (12):
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - Guizhou Provincial People's Hospital, Guiyang
  - Shandong Provincial Hospital, Jinan
  - Zhongda Hospital Southeast University, Nanjing
  - Renmin Hospital of Wuhan University, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - The First Affiliated Hospital of Xi'An Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Henan Provincial People's Hospital, Zhengzhou
- Finland (3):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Hopital Louis Mourier, Colombes, France
- Germany (2):
  - Klinikum Coburg, Coburg
  - University Hospital Münster, Münster
- St. Vincent's University Hospital, Dublin, Ireland
- San Raffaele Hospital, Milan, Italy
- New Zealand (6):
  - Auckland City Hospital, Grafton, Auckland
  - Auckland Hospital DCCM, Auckland
  - Christchurch Hospital, Christchurch
  - Hawke's Bay Hospital, Hastings
  - Rotorua Hospital, Rotorua
  - Wellington Hospital, Wellington
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland
- United Kingdom (8):
  - Stoke Mandeville Hospital, Aylesbury
  - Wycombe General Hospital, High Wycombe
  - Leeds Teaching Hospital, Leeds
  - Lewisham Hospital, London
  - King's College Hospital, London
  - Guy's and St. Thomas Hospital, London
  - Nottingham University Hospital, Nottingham
  - Princess Royal University Hospital, Orpington

REFERENCES:
- [Derived] McCoy IE, Liu KD, Ghamarian E, Quenot JP, Zarbock A, Bihorac A, Khoo B, Gallagher MP, Du B, Joannidis M, Kashani K, Tolwani A, Bagshaw SM, Wald R; STandard versus Accelerated initiation of Renal Replacement Therapy in AKI (STARRT-AKI) Investigators. Dialysis Dependence in Standard versus Accelerated Initiation of KRT in AKI: A Post Hoc Analysis. Clin J Am Soc Nephrol. 2025 May 1;20(5):601-607. doi: 10.2215/CJN.0000000672. Epub 2025 Mar 11. PMID 40232884
- [Derived] Zampieri FG, Serpa-Neto A, Wald R, Bellomo R, Bagshaw SM; STARRT-AKI and RENAL Investigators. Hierarchical endpoints in critical care: A post-hoc exploratory analysis of the standard versus accelerated initiation of renal-replacement therapy in acute kidney injury and the intensity of continuous renal-replacement therapy in critically ill patients trials. J Crit Care. 2024 Aug;82:154767. doi: 10.1016/j.jcrc.2024.154767. Epub 2024 Mar 11. PMID 38461657
- [Derived] Vaara ST, Serpa Neto A, Bellomo R, Adhikari NKJ, Dreyfuss D, Gallagher M, Gaudry S, Hoste E, Joannidis M, Pettila V, Wang AY, Kashani K, Wald R, Bagshaw SM, Ostermann M; STandard vs. Accelerated initiation of Renal Replacement Therapy in Acute Kidney Injury (STARRT-AKI) Investigators. Regional Practice Variation and Outcomes in the Standard Versus Accelerated Initiation of Renal Replacement Therapy in Acute Kidney Injury (STARRT-AKI) Trial: A Post Hoc Secondary Analysis. Crit Care Explor. 2024 Feb 19;6(2):e1053. doi: 10.1097/CCE.0000000000001053. eCollection 2024 Feb. PMID 38380940
- [Derived] Wald R, Kirkham B, daCosta BR, Ghamarian E, Adhikari NKJ, Beaubien-Souligny W, Bellomo R, Gallagher MP, Goldstein S, Hoste EAJ, Liu KD, Neyra JA, Ostermann M, Palevsky PM, Schneider A, Vaara ST, Bagshaw SM. Fluid balance and renal replacement therapy initiation strategy: a secondary analysis of the STARRT-AKI trial. Crit Care. 2022 Nov 24;26(1):360. doi: 10.1186/s13054-022-04229-0. PMID 36424662
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787
- [Derived] STARRT-AKI Investigators; Canadian Critical Care Trials Group; Australian and New Zealand Intensive Care Society Clinical Trials Group; United Kingdom Critical Care Research Group; Canadian Nephrology Trials Network; Irish Critical Care Trials Group; Bagshaw SM, Wald R, Adhikari NKJ, Bellomo R, da Costa BR, Dreyfuss D, Du B, Gallagher MP, Gaudry S, Hoste EA, Lamontagne F, Joannidis M, Landoni G, Liu KD, McAuley DF, McGuinness SP, Neyra JA, Nichol AD, Ostermann M, Palevsky PM, Pettila V, Quenot JP, Qiu H, Rochwerg B, Schneider AG, Smith OM, Thome F, Thorpe KE, Vaara S, Weir M, Wang AY, Young P, Zarbock A. Timing of Initiation of Renal-Replacement Therapy in Acute Kidney Injury. N Engl J Med. 2020 Jul 16;383(3):240-251. doi: 10.1056/NEJMoa2000741. PMID 32668114
- [Derived] STARRT-AKI Investigators. Statistical analysis plan for the Standard versus Accelerated Initiation of Renal Replacement Therapy in Acute Kidney Injury (STARRT-AKI) trial. Crit Care Resusc. 2019 Sep;21(3):162-170. PMID 31462203
- [Derived] STARRT-AKI Investigators. STandard versus Accelerated initiation of Renal Replacement Therapy in Acute Kidney Injury: Study Protocol for a Multi-National, Multi-Center, Randomized Controlled Trial. Can J Kidney Health Dis. 2019 Jun 10;6:2054358119852937. doi: 10.1177/2054358119852937. eCollection 2019. PMID 31218013

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard RRT Initiation: RRT initiation will be guided by the presence of one or more clinical indications. Even in the absence of one of these indications, RRT may be commenced at the discretion of the treating physician.
  Standard RRT initiation: In the absence of kidney function recovery, the initiation of RRT will be permitted if one of the following develops:
  serum potassium ≥ 6.0 mmol/L; pH ≤ 7.20 or serum bicarbonate ≤ 12 mmol/L; evidence of severe respiratory failure, based on a PaO2/FiO2 ≤ 200 and clinical perception of volume overload; and/or persistent AKI > 72 hours following the time of randomization.
Period: Overall Study
Arm/Group | Standard RRT Initiation | Accelerated RRT Initiation
Started | 1507 | 1512
Withdrew Consent | 18 | 9
Randomized Non-eligible | 19 | 31
Lost to Follow-up | 8 | 7
Completed | 1462 | 1465
Not Completed | 45 | 47

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard RRT Initiation | Accelerated RRT Initiation | Total
Number analyzed (Participants) | 1462 | 1465 | 2927
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (13.3) | 64.5 (14.2) | 64.5 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 467 | 470 | 937
  Male | 995 | 995 | 1990
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  North America | 497 | 497 | 994
  Europe | 572 | 574 | 1146
  New Zealand | 80 | 82 | 162
  Brazil | 4 | 4 | 8
  China | 111 | 115 | 226
  Australia | 198 | 193 | 391
Weight - kg [Mean (Standard Deviation); unit: kg] — Population: Number analyzed differs from number enrolled due to missing data.
  kg | 87.9 (25.1) | 87.8 (26.6) | 87.8 (25.8)
Serum creatinine - mg/dl [Mean (Standard Deviation); unit: mg/dl] | 1.3 (1.0) | 1.4 (1.0) | 1.3 (1.0)
Estimated glomerular filtration rate - ml/min/1.73 m2 [Mean (Standard Deviation); unit: ml/min/1.73 m2] | 67.3 (29.8) | 66.0 (29.8) | 66.7 (29.8)
Preexisting conditions - no./total no. (%) - Chronic kidney disease [Count of Participants; unit: Participants] | 626 | 658 | 1284
Preexisting conditions - no./total no. (%) - Hypertension [Count of Participants; unit: Participants] | 823 | 814 | 1637
Preexisting conditions - no./total no. (%) - Diabetes mellitus [Count of Participants; unit: Participants] — Population: Data for this variable was missing for one participant in the standard arm.
  Participants
    number analyzed (Participants) | 1461 | 1465 | 2926
    (all) | 459 | 439 | 898
Preexisting conditions - no./total no. (%) - Heart failure [Count of Participants; unit: Participants] — Population: Data for this variable was missing for one participant in the standard arm.
  Participants
    number analyzed (Participants) | 1461 | 1465 | 2926
    (all) | 204 | 204 | 408
Preexisting conditions - no./total no. (%) - Coronary artery disease [Count of Participants; unit: Participants] — Population: Data for this variable was missing for one participant in the standard arm.
  Participants
    number analyzed (Participants) | 1461 | 1465 | 2926
    (all) | 328 | 320 | 648
Preexisting conditions - no./total no. (%) - Liver disease [Count of Participants; unit: Participants] — Population: Data for this variable was missing for one participant in the standard arm.
  Participants
    number analyzed (Participants) | 1461 | 1465 | 2926
    (all) | 165 | 172 | 337
Preexisting conditions - no./total no. (%) - Metastatic cancer [Count of Participants; unit: Participants] | 84 | 77 | 161
Preexisting conditions - no./total no. (%) - Hematologic cancer [Count of Participants; unit: Participants] | 83 | 87 | 170
Preexisting conditions - no./total no. (%) - HIV infection or AIDS [Count of Participants; unit: Participants] | 13 | 13 | 26
Admission category - no. (%) - Scheduled surgery [Count of Participants; unit: Participants] | 184 | 207 | 391
Admission category - no. (%) - Unscheduled surgery [Count of Participants; unit: Participants] | 289 | 285 | 574
Admission category - no. (%) - Medical [Count of Participants; unit: Participants] | 989 | 973 | 1962
Hospital-acquired risk factor for AKI in previous wk - no./total no. (%) - Cardiopulmonary bypass [Count of Participants; unit: Participants] | 118 | 112 | 230
Hospital-acquired risk factor for AKI in previous wk - no./total no. (%) - Aortic aneurysm repair [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 1461 | 1465 | 2926
    (all) | 74 | 71 | 145
Hospital-acquired risk factor for AKI in previous wk - no./total no. (%) - Other vascular surgery [Count of Participants; unit: Participants] | 77 | 76 | 153
Hospital-acquired risk factor for AKI in previous wk - no./total no. (%) - Major trauma [Count of Participants; unit: Participants] | 55 | 62 | 117
Hospital-acquired risk factor for AKI in previous wk - no./total no. (%) - Obstetric complication [Count of Participants; unit: Participants] | 5 | 5 | 10
Hospital-acquired risk factor AKI previous wk (no./total no. (%)) - Exposure radiocontrast material [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 1460 | 1463 | 2923
    (all) | 375 | 382 | 757
Hospital-acquired risk factor for AKI in previous wk - no./total no. (%) - Receipt of aminoglycoside [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 1458 | 1463 | 2921
    (all) | 148 | 154 | 302
Hospital-acquired risk factor for AKI in previous wk - no./total no. (%) - Receipt of amphotericin B [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 1460 | 1464 | 2924
    (all) | 12 | 9 | 21
Clinical condition at randomization - Sepsis - no. (%) [Count of Participants; unit: Participants] | 834 | 855 | 1689
Clinical condition at randomization - Septic shock - no. (%) [Count of Participants; unit: Participants] | 643 | 640 | 1283
Clinical condition at randomization - SAPS II value [Mean (Standard Deviation); unit: units on a scale] — Results for the Simplified Acute Physiology Score (SAPS) II range from 0 to 163, with higher scores indicating more severe disease and a higher risk of death.
  units on a scale | 59.4 (17.4) | 58.1 (17.4) | 58.8 (17.4)
Clinical condition at randomization - SOFA score [Mean (Standard Deviation); unit: SOFA score (0-24)] — Scores on the Sequential Organ Failure Assessment (SOFA) range from 0 to 24, with higher scores indicating more severe disease and a higher risk of death
  SOFA score (0-24) | 11.8 (3.6) | 11.6 (3.6) | 11.7 (3.6)
Clinical condition at randomization - Mechanical ventilation - no. (%) [Count of Participants; unit: Participants] | 1148 | 1103 | 2251
Clinical condition at randomization - Vasoactive support - no. (%) [Count of Participants; unit: Participants] | 1052 | 1008 | 2060
Clinical condition at randomization - Serum creatinine - mg/dl [Mean (Standard Deviation); unit: mg/dl] — At baseline, the serum creatinine level was defined as the most recent outpatient level obtained during the year pre-ceding the current hospitalization. If this value was not available, the lowest serum creatinine level obtained during the current hospitalization was used to establish the baseline.
  This serum creatinine value was obtained at randomization.
  mg/dl | 3.4 (1.6) | 3.6 (1.7) | 3.5 (1.65)
Clinical condition at randomization - Serum potassium - mmol/liter [Mean (Standard Deviation); unit: mmol/liter] | 4.5 (0.8) | 4.5 (0.8) | 4.5 (0.8)
Clinical condition at randomization - Serum bicarbonate - mmol/liter [Mean (Standard Deviation); unit: mmol/liter] | 19.5 (4.5) | 19.7 (4.7) | 19.6 (4.6)
Clinical condition at randomization - Median urinary output (IQR) - ml/24 hr [Mean (Inter-Quartile Range); unit: ml/24 hr] | 478 [187 to 975] | 450 [190 to 945] | 462 [190 to 955]
Clinical condition at randomization- Oliguria or anuria - no./total no. (%) [Count of Participants; unit: Participants] — Population: Missing data
  Participants
    number analyzed (Participants) | 1420 | 1415 | 2835
    (all) | 618 | 647 | 1265
Clinical condition at randomization- Median cumulative fluid balance (IQR) - ml [Mean (Inter-Quartile Range); unit: ml/ 24 hr] | 2819 [836 to 5603] | 2581 [820 to 5362] | 2691.5 [827 to 5514.8]

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality.
Time Frame: 90 days following study randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard RRT Initiation | Accelerated RRT Initiation
Number analyzed (Participants) | 1462 | 1465
Participants | 639 | 643

2. Secondary Outcome: RRT Dependence
Time Frame: 90 days following study randomization.
Reporting Status: Not Posted

3. Secondary Outcome: Composite of Death or RRT Dependence.
Time Frame: 90 days following study randomization.
Reporting Status: Not Posted

4. Secondary Outcome: Measurement of Estimated Glomerular Filtration Rate.
Time Frame: 90 days following study randomization.
Reporting Status: Not Posted

5. Secondary Outcome: Measurement of Albuminuria.
Time Frame: 90 days following study randomization.
Reporting Status: Not Posted

6. Secondary Outcome: Major Adverse Kidney Outcomes.
Description: Defined as death, RRT dependence or sustained reduction in kidney function (defined as eGFR < 75% baseline eGFR).
Time Frame: 90 days following study randomization.
Reporting Status: Not Posted

7. Secondary Outcome: Mechanical Ventilation-free Days.
Time Frame: Measured from randomization through day 28.
Reporting Status: Not Posted

8. Secondary Outcome: Vasoactive Therapy-free Days
Time Frame: Measured from randomization through day 28.
Reporting Status: Not Posted

9. Secondary Outcome: ICU-free Days
Time Frame: Measured from randomization through day 28.
Reporting Status: Not Posted

10. Secondary Outcome: Hospitalization-free Days
Time Frame: Measured from randomization through day 90.
Reporting Status: Not Posted

11. Secondary Outcome: Death in ICU
Time Frame: Measured in-hospital and at day 28.
Reporting Status: Not Posted

12. Secondary Outcome: EuroQoL EQ-5D-5L.
Description: A measure of health-related quality of life and patient utility.
Time Frame: Measured at day 90 and at day 365.
Reporting Status: Not Posted

13. Secondary Outcome: Health Care Costs.
Time Frame: Measured from baseline through day 365.
Reporting Status: Not Posted

14. Secondary Outcome: Composite of Death or RRT Dependence.
Time Frame: Measured at day 365.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, 90 days following study randomization
Description: All-Cause Mortality was pre-specified to be monitored/assessed only in participants who completed the study. AEs and SAEs were reported from the entire randomized population minus those who withdrew consent
Arm/Group | Standard RRT Initiation | Accelerated RRT Initiation
All-Cause Mortality (participants affected / at risk) | 639/1462 | 643/1465
Serious Adverse Events (participants affected / at risk) | 8/1489 | 15/1503
Other Adverse Events (participants affected / at risk) | 245/1489 | 346/1503
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard RRT Initiation (N=1489) | Accelerated RRT Initiation (N=1503)
Arrhythmia during RRT (Cardiac disorders) | 1 (1) | 2 (2)
CVC - associated bloodstream infection (Surgical and medical procedures) | 0 (0) | 1 (1)
Hemorrhage at site of CVC insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Hemothorax following CVC insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Major bleeding (Surgical and medical procedures) | 0 (0) | 1 (1)
Pneumothorax following CVC insertion (Surgical and medical procedures) | 0 (0) | 2 (3)
RRT - associated hypotension (Vascular disorders) | 4 (4) | 5 (5)
Severe hypocalcemia (Ionized calcium < 0.90 mmol/L) (General disorders) | 0 (0) | 1 (1)
Other (General disorders) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard RRT Initiation (N=1489) | Accelerated RRT Initiation (N=1503)
Hypotension (Vascular disorders) | 131 (188) | 83 (112)
Arrhythmia (Cardiac disorders) | 23 (29) | 37 (45)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Bleeding (Surgical and medical procedures) | 5 (5) | 10 (10)
Allergic reaction (Surgical and medical procedures) | 1 (1) | 1 (1)
Decreased phosphate (<0.5 mmol/liter) (General disorders) | 62 (68) | 112 (124)
Decreased potassium (<3.0 mmol/liter) (General disorders) | 34 (40) | 34 (43)
Decreased ionized calcium (<0.90 mmol/ liter) (General disorders) | 66 (80) | 80 (102)
Pneumothorax or hemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Thrombus (as confirmed on ultrasonography) (Vascular disorders) | 5 (5) | 3 (3)
Arterial puncture (Surgical and medical procedures) | 2 (2) | 3 (3)
Bloodstream infection (Infections and infestations) | 1 (1) | 7 (7)
Other (General disorders) | 19 (20) | 21 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol (2015-10-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT02568722/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT02568722/SAP_001.pdf
  • Informed Consent Form (2016-02-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT02568722/ICF_002.pdf